CLINICAL TRIAL: NCT03756480
Title: Prospective Clinical Study of the Relationship Between Cancer Driving Mutations Found in Endometriotic Implants and the Development of Progesterone Resistance
Brief Title: Cancer Driving Mutations in Endometriosis Lesions and Development of Progesterone Resistance
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00188129; R01HD096147 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis; Endometrial Diseases
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis; Uterine Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial tissue from ectopic and eutopic sites and blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Clinical or surgical diagnosis of Endometriosis, patients undergoing surgical management
  100 participants
- Control Group: No diagnosis of Endometriosis, Patients undergoing Laparoscopic Tubal Ligation
  35 participants

SUMMARY:
This study will test the hypothesis that the molecular changes present in ectopic endometriosis lesions correlate with progesterone-resistant disease (using the criteria defined in this study) and are present in matched eutopic endometrium.

DETAILED DESCRIPTION:
Tissues from 100 patients with endometriosis will be analyzed with droplet digital PCR (ddPCR) targeted sequencing and responders (n=50) will be compared to non-responders (n=50) after controlling confounding factors.

From a subset of the 100 cases, whole exome sequencing (WES) and Methylation-Specific PCR (MSP)-based methylation profiling on microdissected epithelium and stroma will be performed in matched eutopic and ectopic tissues from 20 patients with known cancer-associated mutations or 20 controls.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Gender: female.
* Age: 18-45 years at the time of signing consent.
* Clinical or surgical diagnosis of endometriosis undergoing laparoscopy.
* Controls may not have clinical or surgical diagnosis of endometriosis.
* Regular menstrual cycles.
* BMI between 18-40 kg/m2.
* Sexually active or have had a previous vaginal exam that used a speculum.
* English speaking

Exclusion Criteria:

* Use of any kind of steroidal therapy including oral contraceptives, Norplant, estrogen replacement/supplemental therapy, androgens (Danazol, Cyclomen, Danocrine, testosterone) or progesterone. She may not be taking or be on Celebrex.
* Pregnant.
* Presence of pelvic infection.
* Mullerian anomalies with absence of a cervix.
* History of cancer of the reproductive tract.
* Presence of undiagnosed uterine bleeding.
* Treatment with intrauterine device (IUD) or progestin-containing intrauterine device.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women between the ages of 18-45 undergoing surgical management for endometriosis as cases and women between ages of 18-45 years undergoing elective tubal ligation and no diagnosis of endometriosis.
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of somatic cancer driver mutations in progesterone-resistant versus progesterone-sensitive endometriosis lesions. | Six month
  Digital droplet PCR will be used to identify somatic cancer-driver mutations with the presence of at least one of KRAS or ARID1A or PIK3CA or PPP2R1A cancer-driver mutations to assess any difference between progesterone-resistant endometriosis and progesterone-sensitive endometriosis.

SECONDARY OUTCOMES:
Number of cancer driver mutations in eutopic versus ectopic endometrial tissue in control versus diseased subjects | Six month
  Whole exome sequencing in a subset of patients with progesterone-resistant disease and controls will be done using TruSeq Amplicon Cancer Panel (Illumina) to assess the number of cancer driver mutations.
Difference in DNA methylation PCR profile of endometriotic lesions in ectopic versus eutopic endometrium in control versus diseased subjects. | One month
  DNA methylation profile of eutopic and ectopic endometrial tissue for cases and controls will be done using Raw Illumina 450K methylation array to assess for any difference.

CONTACTS AND LOCATIONS:
Overall Officials: James Segars, MD, FACOG, Principal Investigator — Professor
Locations (3):
- United States (3):
  - Yale School of Medicine, New Haven, Connecticut
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No